CLINICAL TRIAL: NCT01113671
Title: Evaluating the Effect of Vitamin E Treatment on HDL Function of Type 2 Diabetic Patients and the Correlation to Hp Phenotype. A Prospective, Double Blind, Randomized, Placebo Controlled Trial (IDEAL2 Study)
Brief Title: Type 2 Diabetes Haptoglobin Phenotype and Vitamin E
Acronym: IDEAL2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Technion, Israel Institute of Technology (Other)
Responsible Party: Dr. Shany Blum, Laboratory of Vascular Medicine, Faculty of Medicine, Technion - Israel Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HDL005
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus type 2; Haptoglobin phenotype; Vitamin E
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- d-alpha-tocopheryl acetate (Experimental)
  Interventions: Drug: Vitamin E (d-alpha-tocopheryl acetate)

INTERVENTIONS:
Drug: Vitamin E (d-alpha-tocopheryl acetate) — 100% natural source d-alpha-tocopheryl acetate in a soft gel cap
  Arms: d-alpha-tocopheryl acetate
Drug: Placebo — includes inactive Ingredients
  Arms: Placebo

SUMMARY:
This is a biomarker exploratory study which is designed to investigate the function and oxidation of the high density lipoprotein (HDL) (the good cholesterol) in patients with type 2 diabetes mellitus treated with Vitamin E versus placebo and segregated by the type of the Haptoglobin protein they have in their blood.

DETAILED DESCRIPTION:
There exists ample evidence supporting the hypothesis that vitamin E supplementation to Hp 2-2 DM individuals will reduce the incidence of stroke, myocardial infarction and cardiovascular death. Data regarding the association between the Hp 1-1 and 2-1 phenotypes and vitamin E treatment on cardiovascular outcomes such as MI, stroke and CV death is lacking. Furthermore there is no data correlating Hp phenotype, vitamin E and HDL function, structure and oxidation. We wish to evaluate the effect of vitamin E treatment on all diabetic patients with type 2 diabetes on HDL function, structure and oxidation and correlate these parameters to Hp phenotype.

This study will be the first study to prospectively evaluate the interaction of the Hp phenotype and vitamin E in type 2 diabetic patients. As such we wish to evaluate the surrogate marker of reverse cholesterol transport as evidence to the function or dysfunction of the HDL in a relatively small scale study before engaging in a large scale clinical outcome study.

Study objectives. To evaluate the effect of vitamin E treatment on HDL function of reverse cholesterol transport.

Test product. Natural Source Vitamin E (d-α-tocopherol) 400IU administered P.O. as soft gel capsules.

Study population. The study population will be comprised of men and women, age 55 and above with type 2 DM. 90 DM individuals will comprise the treatment phase of the study and will be divided into 30 patients in each Hp phenotype (1-1, 2-1, 2-2).

All 90 patients will be randomized in a double blind fashion into two treatment groups, Vitamin E Natural source 400IU per day versus matching placebo assuring that there will be an equal amount of patients of each phenotype allocated to placebo and Vitamin E.

Study power Calculation_We have calculated that a sample of a total 90 patient (30 in each phenotype) will be required to identify a 30% difference in Reverse Cholesterol Transport between the groups and a statistically significant interaction between phenotype and treatment, with an 80% power and a two sided p value of <0.05.

Study administration. Eligible patients will be identified using the ICARE study database with the help of the ICARE study coordinator at Clalit Health Services. We will identify patients from the 3 Hp phenotypes (those patients were Hp typed as part of the ICARE study and their Hp type is on file). We will then call the patients and they will be asked questions according to the screening questioner to be identified as eligible according to inclusion/exclusion criteria. Those eligible will be invited to the Technion faculty of medicine and will be then recruited to the study after they agree and sign the Informed Consent Form (ICF). Patients will give a blood sample of 50cc of blood at enrollment which will serve as baseline for testing reverse cholesterol transport as well as HDL structure and oxidation. Patients will then be randomized to vitamin E or placebo in a double blinded manner. We will recruit consecutive eligible patients from the ICARE registry till we reach the number of 30 patients in each phenotype and a total of 90 patients. For all 90 treated patients Blood tests (50cc of blood) will be performed after 3 months of treatment, then cross over for an additional 3 months of treatment which in its end the last blood test will be performed (again 50cc). Patients who participate in the treatment phase of the study will have to arrive at the clinic 3 times (baseline and randomization visit, end of first treatment visit and end of second treatment visit).

Analysis. Reverse cholesterol transport results will be compared within and between the groups using paired and unpaired student's t-tests as appropriate. The p for interaction between the 3 phenotype groups and treatment will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 55 and above.
2. Ability to communicate and comply with all study requirements.
3. Able to understand content of informed consent, and has provided written informed consent.
4. Do not take any antioxidant vitamin or drugs including vitamin E, also including all kind of herbal medicines or homeopathic medicine, patients taking such drugs will have to agree to withdrawal from the drug and will be eligible for recruitment after one month of washout.

Exclusion Criteria:

1. Known allergy to vitamin E.
2. Active cardiovascular disease (active stable/unstable angina, less then one year post MI or stroke prior to randomization).
3. Hematological (hemoglobin <10 g/dL), hepatic (aspartate aminotransferase or alanine aminotransferase values >2 x upper limit of normal), or renal disease (serum creatinine >2.5 mg/dL) at baseline.
4. Platelet count <100,000 mm3 and/or abnormal prothrombin or partial thromboplastin time at baseline.
5. Active inflammatory conditions which are likely to require intervention during the course of the study or are regarded as clinically meaningful by the investigator.
6. Active and or treated malignancies within 12 months prior to randomization with the exception of basal cell or squamous cell carcinoma.
7. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
8. Recent history of (within past 12 months) alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1.5 oz distilled spirits).
9. Female subjects who are not either post-menopausal for one year or surgically sterile, and who are not using effective contraceptive methods such as barrier method with spermicidal or an intra-uterine device.
10. History of noncompliance to medical regimens, or subjects unwilling to comply with the study protocol.
11. Administration of any antioxidant vitamins or drugs including vitamin E and not willing to withdrawal and washout for one month prior to enrollment.
12. Administration of any investigational drug within 30 days of planned enrollment into this study.

    * criteria 3,4 will be determined using latest blood tests done in the health plan by the primary physician, patients will be asked to supply those results.

      * all other criteria will be assessed based on patient telephone interview.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Reverse Cholesterol transport of the HDL | 3 months
  Reverse Cholesterol transport of the HDL will be assessed using patients' serum samples in a specified in vitro laboratory assay on baseline, after the first treatment and after the second treatment, Vitamin E treatment effect on this molecular marker will be compared between the 3 different Haptoglobin phenotype patients groups.

SECONDARY OUTCOMES:
HDL oxidation | 3 months
  HDL oxidation will be assessed using patients' serum samples in a specified in vitro laboratory assay on baseline, after the first treatment and after the second treatment, Vitamin E treatment effect on this molecular marker will be compared between the 3 different Haptoglobin phenotype patients groups.
HDL structure | 3 months
  HDL structure will be assessed using patients' serum samples in a specified in vitro laboratory assay on baseline, after the first treatment and after the second treatment, Vitamin E treatment effect on this molecular marker will be compared between the 3 different Haptoglobin phenotype patients groups.
Serum inflammatory markers | 3 months
  Serum inflammatory markers will be assessed using patients' serum samples in a specified in vitro laboratory assay on baseline, after the first treatment and after the second treatment, Vitamin E treatment effect on these molecular markers will be compared between the 3 different Haptoglobin phenotype patients groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, MD PhD, Study Director — Technion, Israel Institute of Technology; Andrew Levy, MD PhD, Study Chair — Technion, Israel Institute of Technology
Locations (1):
- Laboratory of Vascular Medicine, Technion Faculty of Medicine, Haifa, Israel

REFERENCES:
- [Derived] Farbstein D, Blum S, Pollak M, Asaf R, Viener HL, Lache O, Asleh R, Miller-Lotan R, Barkay I, Star M, Schwartz A, Kalet-Littman S, Ozeri D, Vaya J, Tavori H, Vardi M, Laor A, Bucher SE, Anbinder Y, Moskovich D, Abbas N, Perry N, Levy Y, Levy AP. Vitamin E therapy results in a reduction in HDL function in individuals with diabetes and the haptoglobin 2-1 genotype. Atherosclerosis. 2011 Nov;219(1):240-4. doi: 10.1016/j.atherosclerosis.2011.06.005. Epub 2011 Jun 13. PMID 21722898